CLINICAL TRIAL: NCT05245461
Title: Comparison of Patients Who Had Remnant-Preserving Anterior Cruciate Ligament Reconstruction With Healthy Controls In Terms of Muscle Strength and Proprioception
Brief Title: Comparison of Remnant-Preserving Anterior Cruciate Ligament Reconstruction With Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other); Marmara University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK 2021/25
Record Dates: First submitted 2022-02-06; First posted 2022-02-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior Cruciate Ligament Reconstruction: Patients who had remnant-preserving anterior cruciate ligament reconstruction
  Interventions: Other: Assessments
- Healthy Group: People who had no knee surgery or injury
  Interventions: Other: Assessments

INTERVENTIONS:
Other: Assessments — Muscle Strength, Proprioception, Kinesiophobia

SUMMARY:
Anterior cruciate ligament reconstruction stabilizes the knee joint biomechanically and returns the patients back to the sportive activities. Numerous techniques exist to perform an anterior cruciate ligament reconstruction surgery. Remnant- preserving reconstruction technique is performed to increase surgery success rates and to accelerate the post-surgical return to sport process. In general, there is no consensus regarding the clinical outcomes of remnant-preserving anterior ligament reconstruction over standart procedure. The purpose of this study is to compare the patients who had remnant-preserving anterior cruciate ligament reconstruction with healthy controls in terms of muscle strength and proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Anatomical single-bundle ACL reconstruction with AM portal technique using hamstring autograft due to full-thickness ACL tear,
* Endobutton technique was used for femoral fixation,
* Not having any trauma or surgery on the opposite knee,
* Patients with a follow-up period of at least 12 months after surgery.

Exclusion Criteria:

* Fracture of lower extremity accompanying anterior cruciate ligament tear; posterior cruciate ligament, inner and outer lateral ligament tears,
* Patients who have undergone previous surgery on the knee to be evaluated,
* Cases with repeated anterior cruciate ligament reconstruction,
* Having a history of knee joint arthritis (osteoarthritis, inflammatory arthritis),
* Cases with neurological disease will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients who had remnant-preserving ACL reconstruction and healthy controls
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Isokinetic muscle strength | 1 day
  Isokinetic muscle strength values of the Quadriceps Femoris and Hamstring muscles in the knee joint will be measured using the Biodex® System Pro 4 (Biodex Cor. Shirley NY, USA) device. Subjects will perform a warm-up exercise for the knee joint at 75 pedal cycles per minute for three minutes on a bicycle ergometer prior to testing. After the warm-up exercises, the subjects will be allowed to rest for 10 minutes. Subjects will be seated on the isokinetic device chair with their backs perpendicular to 90º. Concentric isokinetic muscle strength measurements of the affected side and unaffected side quadriceps femoris and hamstring muscles of the subjects will be performed with 5 repetitions at 180º /sec, 240º /sec, 300º /sec after the torso, pelvic and thigh belts are attached. Between tests, subjects will be allowed to rest for one minute each. The peak torque values of the cases will be recorded in Nm.
Proprioception | 1 day
  Biodex® System Pro 4 (Biodex Cor. Shirley NY, USA) device will be used to evaluate the proprioception sensation of the knee joint. The subjects will be asked to sit on the isokinetic dynamometer device with the knee joint in 90º flexion. The sense of proprioception of the operated and non-operated knees will be measured at three different angles of 20º, 50º and 70º. During the test, the target angle will be displayed by the device and the limb will be held in this position for 10 seconds. Then, returning to the starting point, the subject will be asked to actively find the target angle with eyes closed. The scores will be averaged by repeating the measurements three times for each reference angle. A rest period of 3 minutes will be allowed between different reference angles.

SECONDARY OUTCOMES:
Kinesiophobia | 1 day
  The level of fear of movement of the participants will be evaluated with the Tampa Kinesiophobia Scale which is a 17-item scale developed to measure fear of movement/re-injury. The scale includes parameters of injury/re-injury and fear and avoidance in work-related activities. The scale evaluates fear of movement with a 4-point Likert-type scoring system (1= Strongly disagree, 4= Totally agree). While the total score is determined between 17-68, a higher score means that the fear of movement is greater.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem Mehmet Ali Aydınlar University, Istanbul
  - Marmara University, Istanbul

IPD SHARING:
Plan to Share IPD: No